CLINICAL TRIAL: NCT01003275
Title: Effects of Oral Paricalcitol on Glucose Tolerance, Immune Cell Function, and Oxidative Stress in Stage 3-4 Chronic Kidney Disease
Brief Title: Metabolic Effects of Paricalcitol
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Ian deBoer, Professor, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 35501-D
Record Dates: First submitted 2009-10-26; First posted 2009-10-28 (Estimated); Results first posted 2013-09-27 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic kidney disease; Vitamin D; Paricalcitol; Placebo; Kidney; Renal; Oxidative Stress; Immune cell function; Glucose; Glucose tolerance
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — paricalcitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paricalcitol followed by placebo (Active Comparator): Participants will receive paricalcitol for 8 weeks, then an 8-week wash-out, then placebo for 8 weeks.
  Interventions: Drug: Paricalcitol; Drug: Placebo
- Placebo followed by paricalcitol (Active Comparator): Participants will receive placebo for 8 weeks, then an 8-week wash-out, then paricalcitol for 8 weeks.
  Interventions: Drug: Paricalcitol; Drug: Placebo

INTERVENTIONS:
Drug: Paricalcitol — Two 1 mcg soft gels by mouth daily for 8 weeks
  Other Names: Zemplar
Drug: Placebo — Two soft gels by mouth daily for 8 weeks

SUMMARY:
The purpose of this study is to determine if treatment with paricalcitol, an active form of vitamin D, has beneficial effects on metabolic abnormalities in people with stage 3-4 Chronic Kidney Disease (CKD).

DETAILED DESCRIPTION:
Persons with chronic kidney disease (CKD) are at markedly increased risk of death, particularly from cardiovascular disease (CVD). A number of metabolic abnormalities may contribute to adverse health outcomes in CKD, including glucose intolerance, altered immune cell function, and oxidative stress. Each of these metabolic stressors is a known complication of CKD. Since these metabolic abnormalities are also known to contribute to the pathogenesis of cardiovascular disease, they are important potential therapeutic targets in CKD.

This study will test whether oral paricalcitol, an active form of vitamin D, will improve glucose tolerance, immune cell function, and reduce oxidative stress in people with stage 3-4 chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Estimated glomerular filtration rate of 15-59 mL/min/1.73m2
* Fasting glucose 100-125 mg/dL
* 18 years and older

Exclusion Criteria:

* Diagnosed with diabetes mellitus
* Use of diabetes medications (insulin or oral hypoglycemics)
* Prior dialysis or transplantation
* Planning to leave the area within 6 months
* Participation in another clinical trial within 30 days
* Treatment with paricalcitol, calcitriol, or corticosteroids in the preceding 8 weeks
* Serum calcium more than 10.2 mg/dL
* Pregnancy or breast-feeding
* Change in dose (within 8 weeks) of Fibrates, Niacin, ACE inhibitors, Angiotensin receptor blockers, Thiazide diuretics, Beta-blockers, Cholecalciferol or Ergocalciferol
* Incontinent of urine
* Cancer (other than skin cancer) within 5 years
* Tuberculosis
* Sarcoidosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian H de Boer, MD, MS, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Result] de Boer IH, Sachs M, Hoofnagle AN, Utzschneider KM, Kahn SE, Kestenbaum B, Himmelfarb J. Paricalcitol does not improve glucose metabolism in patients with stage 3-4 chronic kidney disease. Kidney Int. 2013 Feb;83(2):323-30. doi: 10.1038/ki.2012.311. Epub 2012 Aug 22. PMID 22913981

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 2010 through 2011 from Nephrology clinics associated with the University of Washington.
Period: Overall Study
Arm/Group | Paricalcitol Followed by Placebo | Placebo Followed by Paricalcitol
Started | 11 | 11
Completed | 10 | 11
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paricalcitol Followed by Placebo | Placebo Followed by Paricalcitol | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (10.4) | 65.5 (13.1) | 65.8 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 10 | 10 | 20
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Glucose Area Under the Curve (AUC)
Description: Glucose AUC during a 2-hour oral glucose tolerance test
Time Frame: 8 weeks
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg*min/dL
Arm/Group | During Paricalcitol Treatment | During Placebo Treatment
Number analyzed (Participants) | 22 | 22
mg*min/dL | 20817 (1.2) | 21139 (1.2)

ADVERSE EVENTS:
Arm/Group | During/After Paricalcitol | During/After Placebo
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/21
Other Adverse Events (participants affected / at risk) | 10/22 | 7/21
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | During/After Paricalcitol (N=22) | During/After Placebo (N=21)
Hypercalcemia (Endocrine disorders) | 1 (1) | 0 (0)
Elevated serum creatinine (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fistula placement (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Renal artery stent (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dyspnea with palpitations and lightheadedness (Cardiac disorders) | 1 (1) | 0 (0)
Dyspnea (Cardiac disorders) | 1 (1) | 0 (0)
Elevated blood pressure (Cardiac disorders) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Low back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Paresthesias (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gout flare (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fever (Infections and infestations) | 1 (1) | 0 (0)
Common cold (Infections and infestations) | 1 (1) | 3 (3)
Allergies (Infections and infestations) | 0 (0) | 2 (2)
Vertigo (Nervous system disorders) | 1 (1) | 0 (0)
Rash (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cataract surgery (Eye disorders) | 0 (0) | 1 (1)
Skin cancer removal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less